CLINICAL TRIAL: NCT00388037
Title: A Phase II Study of Sunitinib (SU11248; NSC 736511) in Patients With Recurrent Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Carcinoma
Brief Title: Sunitinib Malate in Treating Patients With Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00647; NCI-2014-00647 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IND.185; NCIC CTG IND.185; CAN-NCIC-IND185; I185; NCIC-185 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-185 (Other: CTEP)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Fallopian Tube Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Primary Peritoneal Cavity Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Primary Peritoneal Cavity Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Primary Peritoneal Cavity Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive sunitinib malate PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib; Sutent
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well sunitinib malate works in treating patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer. Sunitinib malate may inhibit the ability of cancers to grow blood vessels, something they need to grow. It may also shrink tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy (response rate) of sunitinib (sunitinib malate) given orally daily in patients with advanced or metastatic previously treated epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.

II. To assess the toxicity of sunitinib in patients with advanced or metastatic previously treated epithelial ovarian, fallopian tube or primary peritoneal carcinoma.

III. To document cancer antigen 125 (CA125) response rate, early objective progression rate, and, if objective responses are observed, response duration.

OUTLINE:

Patients receive sunitinib malate orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed epithelial ovarian, primary fallopian or primary peritoneal cancer
* Patients must have advanced and/or metastatic disease, incurable by standard therapies
* Patients must have received one or two prior chemotherapy regimens (one must have been platinum containing) and may be either platinum sensitive or platinum resistant

  * Nota bene (NB): For the purposes of this trial, switching from one platinum compound to another for reasons of disease progression or failure to respond will be considered a second regimen; as well, the same regimen given as first and second-line therapy is also considered two regimens
* Presence of clinically and/or radiologically documented disease; at least one site of disease must be unidimensionally measurable as follows:

  * X-ray, physical exam >= 20 mm
  * Spiral computed tomography (CT) scan >= 10 mm; N.B.: Most Canadian hospitals have spiral CT scanning equipment
  * Non-spiral CT scan >= 20 mm; N.B.: Most Canadian hospitals have spiral CT scanning equipment

    * All radiology studies must be performed within 21 days prior to registration (within 28 days if negative)
    * Patients with CA125 as only evidence of disease are not eligible
* Patients must have a life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Hormonal therapy: Patients may have had up to one prior hormonal treatment for metastatic disease; patients must be at least 28 days since last dose of hormonal therapy
* Chemotherapy: Patients must have had a minimum of one and up to two prior chemotherapy regimens, one of which must have contained a platinum agent; patients must be at least 28 days since last chemotherapy treatment and must have recovered from toxic effects
* Radiation: Patients may have had prior radiation therapy; a minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study; radiation must have involved < 30% of functioning bone marrow and there must be measurable disease outside the previously irradiated area (patients whose sole site of disease is in a previously irradiated area are ineligible UNLESS there is evidence of progression, or new lesions have been documented, in the irradiated field); (exceptions may be made however, for low dose, palliative radiotherapy); patients must have recovered from any acute toxic effects from radiation prior to registration
* Previous surgery: Previous major surgery is permitted provided that it has been at least 28 days prior to patient registration and that wound healing has occurred
* Granulocytes (absolute granulocyte count [AGC]) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Bilirubin =< upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Calcium =< 3 mmol/L
* Serum creatinine =< ULN or creatinine clearance >= 60 ml/min if creatinine is > ULN

  * Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft formula
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements; it will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the National Cancer Institute of Canada (NCIC) Clinical Trials Group (CTG) study coordinator that such clearance has been obtained, before the trial can commence in that center; a standard consent form for the trial will not be provided; a copy of the initial full board Research Ethics Board (REB) approval and approved consent form must be sent to the central office; the patient must sign the consent form prior to randomization or registration; please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records
* Patients must be accessible for treatment, response assessment and follow-up; patients registered on this trial must be treated and followed at the participating center; this implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial; investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up
* In accordance with NCIC CTG policy, protocol treatment is to begin within 2 working days of patient registration; exceptions may be made however, regarding the washout period timing for prohibited medications

Exclusion Criteria:

* History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for >= 5 years
* Patients with known brain metastases; (a head CT is not necessary to rule out brain metastases, unless there is clinical suspicion of central nervous system [CNS] involvement); patients with known brain metastases will be excluded from this trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational anticancer agents
* Patients who have received prior treatment with any other antiangiogenic agent or multi-targeted tyrosine kinase inhibitors (e.g. bevacizumab, sorafenib, pazopanib, thalidomide, AZD6474, AMG-706, AZD2171, PTK787, vascular endothelial growth factor [VEGF] Trap, etc.) are ineligible
* Patients with any of the following cardiovascular findings are to be excluded:

  * Corrected QT interval (QTc) prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant electrocardiogram (ECG) abnormalities; an ECG must be done within 14 days prior to registration
  * Current or history of class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Patients with prior anthracycline exposure, previous central thoracic radiation that included heart in radiation port, or a history of NYHA class II cardiac function UNLESS

    * They are currently asymptomatic with respect to cardiac function AND
    * Left ventricular ejection fraction (LVEF) as assessed by multi gated acquisition scan (MUGA) at baseline is > lower limit of normal (LLN) of institution; the MUGA must be done within 14 days prior to registration
  * Poorly controlled hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher)
  * Myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
  * History of pulmonary embolism within the past 12 months
  * History of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; Note: Low molecular weight heparin is permitted provided the patient's international normalized ratio (INR) is =< 1.5; INR must be done within 7 days prior to registration
* Patients with bowel obstruction or any condition (e.g. gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets
* Patients with serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements
  * Active uncontrolled infection
  * Any other medical conditions that might be aggravated by treatment
  * Serious or non-healing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
* Use of agents with proarrhythmic potential (terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide) is not permitted during the study
* The concomitant use of certain drugs is prohibited; patients receiving List A drugs below are not eligible unless >= 7 days since last dose before starting sunitinib and no dosing during the trial; patients receiving List B drugs below are not eligible unless >= 12 days since last dose before starting sunitinib and no dosing during the trial

  * List A: inhibitor/substrates - prohibited 7 days before dosing and during study

    * Azole antifungals (ketoconazole, itraconazole, miconazole), verapamil, clarithromycin, human immunodeficiency virus (HIV) protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir), erythromycin, delavirdine, diltiazem
  * List B: inducer/substrates - prohibited 12 days before dosing and during study

    * Rifampin, phenytoin, rifabutin, St. John's wort, carbamazepine, efavirenz, phenobarbital, tipranavir
* Patients with pre-existing hypothyroidism prior to enrollment are ineligible unless they are euthyroid on medication
* Most women enrolled on this study will have had a prior hysterectomy for ovarian cancer; however, the following are exclusions for enrolment on the study:

  * Pregnant or lactating women; (N.B.: all women of childbearing potential must have a negative urine beta-human chorionic gonadotropin (b-HCG) pregnancy test within 7 days prior to registration)
  * Women of childbearing potential who do not agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; (should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately)
* Known HIV-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Biagi, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Sunitinib Malate)
Started | 31
Completed | 30
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 57 [37 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Partial Response or Complete Response) as Per the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Partial response is defined as a 30% decrease in the sum of the longest diameters of the target lesion maintained for at least 4 weeks; complete response is defined as complete disappearance of disease and cancer related symptoms maintained for at least 4 weeks. The 95% confidence interval for response rate will be calculated. The median and range of the duration of response will be assessed.
Time Frame: Up to 3 years
Population: All response evaluable patients
Measure: Number (95% Confidence Interval); unit: percentage of evalubale patients
Arm/Group | Treatment (Sunitinib Malate)
Number analyzed (Participants) | 28
percentage of evalubale patients | 3.6 [0.1 to 18.3]

ADVERSE EVENTS:
Arm/Group | Treatment (Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib Malate) (N=30)
Neuropathy-Sensory (Nervous system disorders) | 1
Dry eye (Eye disorders) | 1
Dizziness (Nervous system disorders) | 2
Cerebrovascular ischemia (Cardiac disorders) | 1
Hypomagnesemia (Investigations) | 1
Death- NOS (General disorders) | 3
Distension/Bloating and Flatulence (Gastrointestinal disorders) | 1
Watery eye (Eye disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pain-abdominal (General disorders) | 3
Hospitalization for Vomiting (Gastrointestinal disorders) | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 1
Renal Obstruction (Renal and urinary disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Sunitinib Malate) (N=30)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 2
Hypertension (Cardiac disorders) | 15
Fatigue (General disorders) | 28
Fever (General disorders) | 3
Insomnia (General disorders) | 10
Rigors/chills (General disorders) | 6
Sweating (General disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Bruising (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4
Hand-foot (Skin and subcutaneous tissue disorders) | 13
Hypopigmentation (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 10
Dermatology - Other (Skin and subcutaneous tissue disorders) | 8
Hot flashes (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 4
Anorexia (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 19
Diarrhea (Gastrointestinal disorders) | 16
Distension (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 18
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 17
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 24
Obstruction, GI Small bowel NOS (Gastrointestinal disorders) | 2
Taste alteration (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 18
GI - Other (Gastrointestinal disorders) | 5
Hemorrhage, GI Rectum (Blood and lymphatic system disorders) | 5
Hemorrhage, GU Vagina (Blood and lymphatic system disorders) | 3
Infection with normal ANC Bladder (Infections and infestations) | 2
Infection with normal ANC Urinary tract NOS (Infections and infestations) | 3
Infection with unknown ANC Upper airway NOS (Infections and infestations) | 2
Edema: head and neck (Blood and lymphatic system disorders) | 5
Edema: limb (Blood and lymphatic system disorders) | 6
Muscle weakness Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 7
Mood alteration Anxiety (Nervous system disorders) | 7
Mood alteration Depression (Nervous system disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 15
Syncope (Nervous system disorders) | 2
Blurred vision (Eye disorders) | 3
Watery eye (Eye disorders) | 7
Ocular - Other (Eye disorders) | 2
Pain Abdomen NOS (General disorders) | 20
Pain Back (General disorders) | 13
Pain Bladder (General disorders) | 2
Pain Extremity-limb (General disorders) | 4
Pain Head/headache (General disorders) | 13
Pain Joint (General disorders) | 6
Pain Muscle (General disorders) | 6
Pain Neck (General disorders) | 2
Pain Oral cavity (General disorders) | 3
Pain Pelvis (General disorders) | 5
Pain Rectum (General disorders) | 2
Pain Throat/pharynx/larynx (General disorders) | 2
Pain - Other (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Incontinence, urinary (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 5
Urine color change (Renal and urinary disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less